CLINICAL TRIAL: NCT05315050
Title: Impact of Menstrual Health Education on Knowledge, Attitudes and Self Care Behavior of Female Adolescents With Primary Dysmenorrhea
Brief Title: Menstrual Health Education's Impact on Knowledge, Attitudes and Self Care Behavior of Dysmenorrheal Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mahrukh Usmani
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Primary Dysmenorrhea
Keywords: Dysmenorrhea; Menstruation; Adolescent; Knowledge; Attitude
MeSH Terms: conditions — Dysmenorrhea; Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational session and Informational Pamphlet (Experimental)
  Interventions: Other: Educational session and Information Pamphlet
- Informational Pamphlet (Active Comparator)
  Interventions: Other: Information Pamphlet

INTERVENTIONS:
Other: Educational session and Information Pamphlet — Each session will last for 50 minutes that will consist on lecturing, discussion about improving adolescent girls' menstrual knowledge, promoting a more positive attitude, encourage confidence, self-care behavior, physical activity and improve pain relief practice.
  Exercise advice: The exercise protocol will include aerobic exercise such as jogging, which perform in the interventional group, three times a week, and for 10 to 30 min.
  Stretching's advice: Piriformis stretching (5 repitition×20seconds), Cobra Pose. (5 repitition×20seconds), Adductor stretching. (5 repitition×20seconds), Sit up (10 repetition × 3 sets), Bridge exercise (10 repetition × 3 sets), Kegel exercise (10repetition × 3 sets), Pelvic eleva¬tion (10repetition × 3 sets), three times a week.
  Arms: Educational session and Informational Pamphlet
Other: Information Pamphlet — Pamphlets consist of information about primary dysmenorrhea its causes, symptoms (onset, duration, location, prognosis) and treatment strategies (taking hot bath, heating pad, yoga, exercise, maintaining hygiene, modifying life style) Emphasized on that menstruation is a not a disease it's a natural life experience.
  Arms: Informational Pamphlet

SUMMARY:
This study will be a randomized controlled trial. This study will be conducted in F G modal for girls' I/8-4, Federal Government College for Women and Islamabad Model College for Girls. A sample size of 138 patients will be taken. Patients will be divided into two groups by lottery method. Group A will receive Educational sessions and informational pamphlet while Group B will only receive the pamphlets. Experimental group will receive for 4 sessions (2 per week). The outcome measures Menstrual Attitude Questionnaire (MAQ), Dysmenorrhoeic Knowledge Scale (DKS) and Dysmenorrhoeic Self-Care behavior Scale (DSCBS) will be measured at baseline, and at the end of week 2 and after 3 months. Data will be analyzed by SPSS 21.

DETAILED DESCRIPTION:
Dysmenorrhea, characterized by painful cramps of the uterus during menstruation. It affects up to 95% of menstruating women. Dysmenorrhea is classified as primary and secondary dysmenorrhea. Primary dysmenorrhea is defined as menstrual cramping pain that occurs immediately before or during menstruation in the absence of any pelvic pathology. The pain commonly starts within 3 years of menarche (the first menstrual period). Prevalence of primary dysmenorrhea varies from between 16 to 91% in reproductive aged women. Primary dysmenorrhea is the leading women hood problem that affects 90% of adolescent girls. Its prevalence decreases with increasing age in a large percentage of sufferers.

A study conducted in China concluded that nurse-managed education program improved adolescent girls' menstrual knowledge, promoted a more positive attitude, encouraged confidence, and improved pain relief practice. Another study conducted in Taiwan showed that the prevalence in dysmenorrhea in female adolescents was high, but they were lacking in dysmenorrhea related self-care knowledge. An Australian study concluded that the prevalence and impact of dysmenorrhea on Grade 11 and 12 girls is high, girls need more education on this area to prevent unnecessary suffering and interruption to school routine as they lack knowledge of and experience with effective treatment. A cross-sectional, internet-based survey was conducted, concluded that one in 3 women quit daily activities owing to menstrual symptoms. Half of all women did not mention menstrual complaints being the reason for transferring tasks in a family setting. However, considering the impact of menstrual symptoms on daily activities in a large group of women, it is time to open the societal dialogue and improve education for both patients and doctors.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent girls aged 13-19 years of age.
* Experienced dysmenorrhea cramps 2 or more times during the last 6 months.
* Dysmenorrhea diagnosed using working ability, location, intensity, days of pain, dysmenorrhea (WaLIDD) score.

Exclusion Criteria:

* • Unwilling to participate.

  * Known cases of depression, anxiety, bipolar disorder, and other mood disorder
  * Minors whose parents do not allow.

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 138 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Menstrual Attitude Questionnaire (MAQ) | 3 months
  This scale was originally developed by Brooks-Gunn and Ruble and modified by Li. It consists of 32 items with five dimensions, including menstruation as a debilitating event, menstruation as a bothersome event, menstruation as a natural event, anticipation and prediction of the onset of menstruation, and denial of any effect of menstruation. Each item is scored on a 7-point Likert scale from 1 (disagree strongly) to 7 (agree strongly). Total scores range from 32 to 224, with the higher score representing a more positive attitude toward menstruation.
Dysmenorrhoeic Knowledge Scale (DKS) | 3 months
  The DKS was designed based on the researchers' clinical experiences and previous studies. The scale included 20 questions with yes/no answers. If the subject answered correctly, it was rated as 1; if answered incorrectly, it was rated as 0. Total scores ranged from 0 to 20 with the higher score representing a better knowledge of dysmenorrhea
Dysmenorrhoeic Self-Care behavior Scale (DSCBS) | 3 months
  This scale was designed based on the researchers' clinical experiences and previous literature. It contains 22 items. Each item is scored on a 4-point Likert scale from 0 (never) to 3 (always). Total scores ranged from 0 to 66, with the higher score representing a more positive self-care behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Hadia Nadeem, M.Phil PT, Principal Investigator — Riphah International University
Locations (1):
- Islamabad Model College for Girls, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No